CLINICAL TRIAL: NCT03734484
Title: Gram Type Infection-Specific Sepsis Identification Using Machine Learning
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: study was not started.
Sponsor: Dascena (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 01072019
Record Dates: First submitted 2018-11-01; First posted 2018-11-08 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Sepsis; Severe Sepsis; Septic Shock
Keywords: Dascena; Gram infection; antibiotic administration; machine learning; algorithm; diagnostic
MeSH Terms: conditions — Sepsis; Shock, Septic; Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gram type infection-specific algorithm (Experimental): The experimental arm will involve patients monitored by the Gram type infection-customized version of InSight.
  Interventions: Diagnostic Test: InSight
- Standard treatment protocol (No Intervention): The control arm will involve patients treated with the regular diagnosis and treatment protocol for gram-type infection, where fluid cultures are run to determine infection type.

INTERVENTIONS:
Diagnostic Test: InSight — The InSight algorithm which draws information from a patient's electronic health record (EHR) to predict the onset of severe sepsis, and in this study will be customized to differentiate between various Gram-type infections.
  Arms: Gram type infection-specific algorithm

SUMMARY:
The focus of this study will be to conduct a prospective, randomized controlled trial (RCT) at Cape Regional Medical Center (CRMC), Oroville Hospital (OH), and UCSF Medical Center (UCSF) in which a Gram type infection-specific algorithm will be applied to EHR data for the detection of severe sepsis. For patients determined to have a high risk of severe sepsis, the algorithm will generate automated voice, telephone notification to nursing staff at CRMC, OH, and UCSF. The algorithm's performance will be measured by analysis of the primary endpoint, time to antibiotic administration. The secondary endpoint will be reduction in the administration of unnecessary antibiotics, which includes reductions in secondary antibiotics and reductions in total time on antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* All adults above age 18 who are a member of one of the three subpopulations studied in this trial (patients with Gram-positive infection, patients with Gram-negative infection, and patients with mixed Gram-positive and Gram-negative infection) are eligible to participate in the study.

Exclusion Criteria:

* Under age 18
* No record of Gram infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in time to antibiotic administration | Through study completion, an average of 8 months
  Change in time period between diagnosis of Gram infection and administration of antibiotics to treat infection

SECONDARY OUTCOMES:
Change in administration of unnecessary antibiotics | Through study completion, an average of 8 months
  Changes in amount of secondary antibiotics administered
Change in administration of unnecessary antibiotics | Through study completion, an average of 8 months
  Changes in total hours spent on antibiotics

CONTACTS AND LOCATIONS:
Overall Officials: Ritankar Das, MSc, Principal Investigator — Dascena

REFERENCES:
- [Background] Calvert J, Mao Q, Hoffman JL, Jay M, Desautels T, Mohamadlou H, Chettipally U, Das R. Using electronic health record collected clinical variables to predict medical intensive care unit mortality. Ann Med Surg (Lond). 2016 Sep 6;11:52-57. doi: 10.1016/j.amsu.2016.09.002. eCollection 2016 Nov. PMID 27699003
- [Background] Shimabukuro DW, Barton CW, Feldman MD, Mataraso SJ, Das R. Effect of a machine learning-based severe sepsis prediction algorithm on patient survival and hospital length of stay: a randomised clinical trial. BMJ Open Respir Res. 2017 Nov 9;4(1):e000234. doi: 10.1136/bmjresp-2017-000234. eCollection 2017. PMID 29435343
- [Background] Mao Q, Jay M, Hoffman JL, Calvert J, Barton C, Shimabukuro D, Shieh L, Chettipally U, Fletcher G, Kerem Y, Zhou Y, Das R. Multicentre validation of a sepsis prediction algorithm using only vital sign data in the emergency department, general ward and ICU. BMJ Open. 2018 Jan 26;8(1):e017833. doi: 10.1136/bmjopen-2017-017833. PMID 29374661